CLINICAL TRIAL: NCT05841147
Title: Reduction of Microembolism After Stent-Assisted Coil Embolization of Unruptured Intracranial Aneurysms by Administration of Tirofiban：A Randomized, Controlled, Double-blind Trial
Brief Title: Reduction of Microembolism After the Intervention Surgery of Intracranial Aneurysms by Administration of Tirofiban
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lu Hua (Other)
Responsible Party: Sponsor-Investigator, Lu Hua, Chief physician, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ANHSI
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Intracranial Aneurysm
Keywords: Aneurysm; Tirofiban; Stent-Assisted Coil Embolization
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm | interventions — Tirofiban; Saline Solution

STUDY DESIGN:
Intervention Model Description: The intervention group: An intravenous bolus (6µg/kg) over a 3 min period and a maintenance dose of 0.1µg/kg/min for 18 hour were used in this group.
  The control group: The same dose of normal saline was used instead of tirofiban.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding all personnel who may interfere with the trial results, such as Participant, Care Provider, Investigator and Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): An intravenous bolus (6µg/kg) over a 3 min period and a maintenance dose of 0.1µg/kg/min for 18 hour were used in this group.
  Interventions: Drug: Tirofiban
- The control group (Active Comparator): The same dose of normal saline was used instead of tirofiban.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Tirofiban — Intravenous administration of tirofiban
  Arms: The intervention group
Drug: normal saline — Intravenous administration of normal saline
  Arms: The control group

SUMMARY:
The goal of this clinical trial is to investigate whether intravenous injection of tilofiban can reduce microembolism in patients with unruptured intracranial aneurysms after Stent-Assisted Coil Embolization.The main questions it aims to answer are:

* Is it safe to inject tirofiban intravenously during interventional treatment of intracranial aneurysms？
* What dose of tirofiban is safe and effective?

DETAILED DESCRIPTION:
We aim to reduce microembolism in patients with unruptured intracranial aneurysms after Stent-Assisted Coil Embolization.

ELIGIBILITY:
Inclusion Criteria:

* Age was between 18 and 75 years old;
* Unruptured aneurysm with surgical indications;
* Stent assisted coil embolization treatment was received ;
* The patient was willing to receive intervention treatment.

Exclusion Criteria:

* Complicated with hemorrhagic cerebrovascular diseases such as cerebral vascular malformations and moyamoya disease or their medical history;
* Recent (within 1 year) bleeding symptoms such as gastrointestinal bleeding, clinically significant urinary/reproductive tract bleeding, and skin blueness;
* Dissecting aneurysm, pseudoaneurysm, and bullous aneurysm;
* A known history of coagulation disorders, platelet abnormalities, or thrombocytopenia; 5. Platelet count less than 150 × 109/L；
* A history of major surgical procedures or severe physical trauma within one month;
* Severe uncontrolled hypertension (systolic blood pressure>160mmHg and/or diastolic blood pressure>100mmHg);
* Hemorrhagic retinopathy;
* Chronic hemodialysis;
* Renal insufficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-25 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Microembolism | Within 72 hours after surgery
  Number of microembolism

SECONDARY OUTCOMES:
The incidence of microembolism | Within 48 hours after surgery
  The incidence of microembolism

OTHER OUTCOMES:
Hemorrhage | Within 48 hours after surgery
  The incidence of Hemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, China